CLINICAL TRIAL: NCT07351461
Title: Quantitative and Qualitative Study of Anxiety in Patients Under Active Surveillance for Localized Prostate Cancer and Their Partners.
Brief Title: Anxiety in Patients Under Active Surveillance for Localized Prostate Cancer and Their Partners.
Acronym: ANCAPRO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2023_0457
Record Dates: First submitted 2025-09-23; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Anxiety
MeSH Terms: conditions — Prostatic Neoplasms; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patient on active surveillance — * First, a quantitative cross-sectional study of patients on active surveillance at Lille University Hospital, which will aim to determine the prevalence of anxiety disorders in patients and, if possible, in their partners.
  * Then, a qualitative study to explore the potential causes of this anxiety.

SUMMARY:
Prostate cancer (PCa) is the most common cancer and the third leading cause of cancer-related death among men in France.

Active surveillance is one of the management options for low-risk prostate cancer. Its aim is to delay or avoid radical treatment, such as surgery or radiotherapy, which can cause side effects including urinary incontinence, erectile dysfunction, or radiation-induced cystitis. Active surveillance involves regular monitoring of potential tumor progression through serum PSA testing, MRI scans, and prostate biopsies.

Few studies have investigated the psychological adjustment of patients undergoing active surveillance for prostate cancer, and even fewer have explored the relationship between the patients' anxiety symptoms and those of their partners. To our knowledge, no study has yet quantitatively or qualitatively assessed the anxiety of both patients and their partners. It appears essential to better characterize the anxiety symptoms in these individuals in order to offer them appropriate psychological support.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients who started active surveillance for localized prostate cancer from 2007 to 2023 and are followed in the Urology Department of Lille University Hospital.
* Affiliation to a social security scheme.
* Obtaining patient consent.
* Having a life partner or an unidentified partner recognized as the person sharing the patient's daily life

Exclusion Criteria:

* Lack of proficiency in the French language.
* Minor patients, those under legal protection measures, or deprived of liberty.
* Lack of medical insurance coverage.
* Patients refusing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients who started active surveillance for localized prostate cancer between 2007 and 2023 and are followed in the Urology Department of Lille University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 432 (Estimated)
Dates: Start 2025-03-23 (Actual); Primary Completion 2027-03-23 (Estimated); Study Completion 2027-03-23 (Estimated)

PRIMARY OUTCOMES:
Prevalence of anxiety symptoms in patients under active surveillance for prostate cancer. | 12 months
  Total score of the 'Memorial Anxiety Scale for Prostate Cancer' questionnaire, whose French translation has been validated (Touzani et al., 2019). Patients scoring >27/54 are classified as anxious.

SECONDARY OUTCOMES:
Prevalence of anxiety symptoms in the partners of patients under active surveillance for prostate cancer | 12 months
  Questionnaire assessing anxiety (STAI-Y questionnaire).
To determine the clinical predictive factors of anxiety in patients on active surveillance. | 12 months
  Use of questionnaires assessing general anxiety (STAI-Y questionnaire) in patients and their partners.
To determine the predictive factors of anxiety in terms of personal and dyadic coping strategies. | 12 months
  Assessment of intra- and interpersonal emotional skills.
To identify the potential causes of anxiety. | 12 months
  Participants scoring between 115 and 145 on the DCI are considered within the normal range. A score below 115 indicates that participants use dyadic coping strategies less frequently than average. A score above 145 indicates that participants use dyadic coping strategies more frequently than average.
Determine the predictive factors of anxiety in terms of interpersonal skills in patients and their partners. | 12 months
  Assessment of intra- and interpersonal emotional skills.
Prevalence of anxiety symptoms in the partners of patients under active surveillance for prostate | 12 months
  Questionnaire assessing the management of emotions (S-PEC questionnaire).
Prevalence of anxiety symptoms in the partners of patients under active surveillance for prostate | 12 months
  Questionnaire assessing the stress (Dyadic coping inventory questionnaire).
To determine the clinical predictive factors of anxiety in patients on active surveillance. | 12 months
  Use of questionnaires assessing the stress (Dyadic coping inventory questionnaire) in patients and their partners.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No